CLINICAL TRIAL: NCT05474638
Title: Comparison of Mechanomyographic 100 Versus 200 Hz 5 Second Tetanic Fade Ratios During Neuromuscular Block Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire UCLouvain Namur (Other)
Responsible Party: Principal Investigator, Philippe Dubois, Professor Philippe Dubois, Centre Hospitalier Universitaire UCLouvain Namur
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TFR 100 vs 200 Hz
Record Dates: First submitted 2022-07-15; First posted 2022-07-26 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Neuromuscular Blockade
Keywords: Residual neuromuscular block; Mechanomyography; Tetanic nerve stimulation
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Intervention Model Description: Controlateral and simultaneous comparison of two different neuromuscular transmission monitorings in a cohort of 20 anesthetised patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controlateral and simultaneous comparison of neuromuscular transmission monitors (Other): Controlateral and simultaneous comparison of responses from acceleromyography- and mechanomyography-based neuromuscular transmission monitors in the same patients.
  Interventions: Device: Isometric Thumb Force (isometric mechanomyography) compared to TOF-Watch SX (acceleromyography)

INTERVENTIONS:
Device: Isometric Thumb Force (isometric mechanomyography) compared to TOF-Watch SX (acceleromyography) — Comparison of mechanomyographic measurements of thumb adduction's force induced by 100 versus 200 Hz 5 seconds tetanic ulnar nerve stimulation during neuromuscular block spontaneous recovery monitored by acceleromyography on the controlateral arm.

SUMMARY:
Two recent pilot studies suggested the potential interest of 100 and 200 Hz tetanic stimulations to detect with mechanomyography (MMG) very low levels of residual neuromuscular blockade (NMB). The Tetanic Fade Ratio (TFR, residual force after 5 seconds / maximal force) measured quantitatively by MMG during tetanic stimulation at 100 or 200 Hz could provide today a more consistent response than the train-of-four (TOF) ratio provided by acceleromyography (AMG) to this search for detection of low levels of residual NMB.

This study was designed to evaluate for the first time in anesthetized patients the evolution of NMB spontaneous recovery with 5-second 100 and 200 Hz tetanic stimulations compared to TOF, and to test the hypothesis that a 200 Hz TFR would better and longer detect low levels of residual paralysis than AMG TOF ratio and 100 Hz TFR.

DETAILED DESCRIPTION:
MATERIALS AND METHODS Patient management The monocentric study protocol was approved before patients' inclusion by the Institutional Ethical Committee (CHU UCL Namur, Yvoir, Belgium, OM 050, under unique belgian registration number B0392022000035).

It was performed in accordance with the ethical standards of the Declaration of Helsinki and was included in the Clinical Trials Registry (XXX).

After obtaining written informed consent from all participants, 20 patients with American Society of Anesthesiologists (ASA) grades I to II (aged 18 to 65 years), who were scheduled to undergo rhinoplasty or rhinoseptoplasty under general anaesthesia, were included in the study. The exclusion criteria were pregnant or breastfeeding women, patients with renal or hepatic insufficiency, patients with neurological disorders, and any patient with a suspected allergy to the drugs used in the protocol or receiving medications that could interfere with neuromuscular transmission. The patient's height, weight, age, and sex were recorded in the protocol to define the population investigated.

The patients were conventionally monitored with a pulse oximeter, a three-lead electrocardiogram and a non-invasive blood pressure monitor scheduled in automatic mode at 5-minute intervals. An intravenous catheter was inserted into their forearm for crystalloid infusion (side at random). Neuromuscular transmission monitoring (NMTM) was set up according to a specific protocol.

Total intravenous anaesthesia was induced with continuous infusion of remifentanil 0.25 µg/kg/min and continuous infusion of propofol 1% to obtain theoretical plasma concentrations ranging from 3 to 6 µg/mL (Diprifusor Cardinal Health, Basingstoke, UK). Lidocaine 1 mg/kg was also given as an intravenous bolus. After loss of consciousness, manual ventilation was provided during NMTM calibration and the initial NMB baseline measurements. Then, rocuronium 0.45 mg/kg was administered. Non-invasive automatic blood pressure measurement was suspended during the neuromuscular onset to avoid dissimilar distribution of the rocuronium in the two arms. Tracheal intubation was performed when the TOF count reached zero. Automatic non-invasive blood pressure measurement was reactivated. Mechanical ventilation (closed circuit, 40% oxygen in air) maintained end-tidal CO2 within the normal range. Anesthesia was maintained with the continuous intravenous administration of remifentanil 0.15 µg/kg/min and propofol with a target plasma concentration of 2 to 4 µg/mL. Blankets prevented heat loss from the body and both arms, and the oropharyngeal temperature was kept stable. Postoperative analgesia was provided with paracetamol, tramadol and alizapride at the end of surgery.

Neuromuscular transmission monitoring

All recordings were performed during general anesthesia. The skin was cleaned with diethyl ether, and two electrodes were placed above the ulnar nerve on each wrist.

A TOF-Watch SX® (Alvesia Pharma, France) (TWSX) was set on the left hand. The accelerometric transducer was taped on the thumb's pulp, and the hand was inserted and held inside an SL TOF tube. Another TOF-Watch® (Organon-Technika, Copenhagen, Denmark) designed to deliver high-frequency tetanic stimulations (including 100 and 200 Hz) was connected to the electrodes on the right arm, which was equipped with an Isometric Thumb Force (ITF®) handgrip designed to record the force (N) of isometric thumb adduction during electrical stimulations. The Visual-ITF® software recorded all measurements for further off-line analysis. Each tetanic signal was described in a 5 sec window starting from the 1 Newton value. If this 1N threshold was not reached, the recording was excluded from the analysis.

Both arms were positioned alongside the body on soft padding to protect nerve structures from any extra focal pressure.

Supra-maximal stimulation and initial calibration were obtained using the TWSX internal automatic sequence, and the current intensity displayed was applied on both sides. Then, TOF stimulations were applied at 15-second intervals during a short stabilisation period. On the TWSX side, four T4/T1 ratios were recorded to determine the initial baseline (mean of four values) before NMBA administration. On the ITF side, two consecutive tetanic stimulations (100 and 200 Hz at random) were applied for 5 seconds, with a two-minute interval to avoid any potentiation. Consecutive TOF stimulations every 15 seconds were applied to monitor the NMB, from the onset and, during surgery, until the spontaneous recovery of a normalized TOF ratio of 0.9 on the TWSX side and even further. Both tetanic stimulations (same order as previously) were applied alternately with 2-minute intervals on several steps of recovery and until recovering 90% of the initial TFR with both stimulation patterns.

Data collection and statistical analysis On the TWSX side, the TOF ratio provided after each 2Hz TOF stimulation was displayed and recorded. We calculated 90% of the initial baseline mean value to determine the normalised TOF ratio 0.9 recovery threshold using the following formula: normalised TOF ratio 0.9 = sum of 4 TOF ratio × 9/40, with the result rounded up.

On the ITF side, a Tetanic Fade Ratio (TFR) was determined to quantify any fade occurring during the muscle contraction: referring to the resting level just before the contraction, the residual force at the end of 5 seconds of stimulation was divided by the maximal force obtained during the contraction to provide a ratio.

Based on a previous pilot study using the same material and the same stimulating patterns, a sample of 20 patients was determined to provide a significant difference between the TFRs recorded with 100 and 200 Hz tetanic stimulations at the time of AMG TOF ratio 0.9 recovery. We expected to have enough power (0.8 at that stage) to detect a significant difference during an additional period of recovery. The alpha error was 0.05.

Off-line data analysis was based on the archived files. Using R software version 3.3.6 (R Project for Statistical Computing, Vienna, Austria), Student's t-tests were performed to compare the TFR obtained after 100- or 200-Hz stimulations at initial baseline and at several classical levels of spontaneous recovery on the TWSX side:

* TOF count 1,
* TOF ratio 0.5,
* TOF ratio 0.9
* Normalized TOF ratio 0.9
* TOF ratio 0.95
* TOF ratio 1.0 Then, both tetanic stimulations were repeated every 5 minutes until TFR reached 0.9 to quantify any further period of analysis of low levels of residual blockade.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* written informed consent
* general anesthesia for rhino(septo)plasty

Exclusion Criteria:

* pregnant or breastfeeding women
* patients with renal or hepatic insufficiency
* patients with neurological disorders
* patients with a suspected allergy to the drugs used in the protocol
* patients receiving medications that could interfere with neuromuscular transmission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
100 vs 200 Hz Tetanic Fade Ratio comparison | During surgery while the neuromuscular block spontaneously recovers from AMG TOF count 1 until TOF ratio 1.0
  To compare 100 and 200 Hz TFR at different literature based spontaneous recovery levels recorded by acceleromyography on the other arm: TOF count 1, TOF ratio 0.5 and TOF ratio 0.9 / normalized 0.9 / 0.95 / 1.0.

SECONDARY OUTCOMES:
Quantification of any remaining MMG fade with 200 Hz stimulation after AMG TOF ratio 0.9 recovery | During surgery while the neuromuscular block spontaneously recovers from AMG TOF ratio 0.9 until MMG 200 Hz TFR > 0.9
  To quantify any significant deeper fade occurring with 200 Hz compared to 100 Hz during further stages of spontaneous recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Alain D'Hollander, Prof, Study Chair — Fondation pour l'Anesthésie-Réanimation, Vaduz
Locations (1):
- CHU Dinant-Godinne, Yvoir, Belgium

REFERENCES:
- [Background] Ali HH, Utting JE, Gray C. Stimulus frequency in the detection of neuromuscular block in humans. Br J Anaesth. 1970 Nov;42(11):967-78. doi: 10.1093/bja/42.11.967. No abstract available. PMID 5488360
- [Background] Gissen AJ, Katz RL. Twitch, tetanus and posttetanic potentiation as indices of nerve-muscle block in man. Anesthesiology. 1969 May;30(5):481-7. doi: 10.1097/00000542-196905000-00001. No abstract available. PMID 4305092
- [Background] Waud BE, Waud DR. The relation between tetanic fade and receptor occlusion in the presence of competitive neuromuscular block. Anesthesiology. 1971 Nov;35(5):456-64. doi: 10.1097/00000542-197111000-00003. No abstract available. PMID 4329144
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Ali HH, Savarese JJ, Lebowitz PW, Ramsey FM. Twitch, tetanus and train-of-four as indices of recovery from nondepolarizing neuromuscular blockade. Anesthesiology. 1981 Apr;54(4):294-7. doi: 10.1097/00000542-198104000-00007. PMID 6452074
- [Background] Stanec A, Heyduk J, Stanec G, Orkin LR. Tetanic fade and post-tetanic tension in the absence of neuromuscular blocking agents in anesthetized man. Anesth Analg. 1978 Jan-Feb;57(1):102-7. doi: 10.1213/00000539-197801000-00019. PMID 204226
- [Background] Kopman AF, Epstein RH, Flashburg MH. Use of 100-Hertz tetanus as an index of recovery from pancuronium-induced non-depolarizing neuromuscular blockade. Anesth Analg. 1982 May;61(5):439-41. PMID 7199868
- [Background] Eikermann M, Vogt FM, Herbstreit F, Vahid-Dastgerdi M, Zenge MO, Ochterbeck C, de Greiff A, Peters J. The predisposition to inspiratory upper airway collapse during partial neuromuscular blockade. Am J Respir Crit Care Med. 2007 Jan 1;175(1):9-15. doi: 10.1164/rccm.200512-1862OC. Epub 2006 Oct 5. PMID 17023729
- [Background] Plaud B, Debaene B, Donati F, Marty J. Residual paralysis after emergence from anesthesia. Anesthesiology. 2010 Apr;112(4):1013-22. doi: 10.1097/ALN.0b013e3181cded07. No abstract available. PMID 20234315
- [Background] Kirmeier E, Eriksson LI, Lewald H, Jonsson Fagerlund M, Hoeft A, Hollmann M, Meistelman C, Hunter JM, Ulm K, Blobner M; POPULAR Contributors. Post-anaesthesia pulmonary complications after use of muscle relaxants (POPULAR): a multicentre, prospective observational study. Lancet Respir Med. 2019 Feb;7(2):129-140. doi: 10.1016/S2213-2600(18)30294-7. Epub 2018 Sep 14. PMID 30224322
- [Background] Blobner M, Hunter JM, Meistelman C, Hoeft A, Hollmann MW, Kirmeier E, Lewald H, Ulm K. Use of a train-of-four ratio of 0.95 versus 0.9 for tracheal extubation: an exploratory analysis of POPULAR data. Br J Anaesth. 2020 Jan;124(1):63-72. doi: 10.1016/j.bja.2019.08.023. Epub 2019 Oct 10. PMID 31607388
- [Background] Capron F, Alla F, Hottier C, Meistelman C, Fuchs-Buder T. Can acceleromyography detect low levels of residual paralysis? A probability approach to detect a mechanomyographic train-of-four ratio of 0.9. Anesthesiology. 2004 May;100(5):1119-24. doi: 10.1097/00000542-200405000-00013. PMID 15114208
- [Background] Suzuki T, Fukano N, Kitajima O, Saeki S, Ogawa S. Normalization of acceleromyographic train-of-four ratio by baseline value for detecting residual neuromuscular block. Br J Anaesth. 2006 Jan;96(1):44-7. doi: 10.1093/bja/aei273. Epub 2005 Nov 18. PMID 16299046
- [Background] Dubois PE, Mitchell J, Regnier M, Passeraub PA, Moreillon F, d'Hollander AA. The interest of 100 versus 200 Hz tetanic stimulations to quantify low levels of residual neuromuscular blockade with mechanomyography: a pilot study. J Clin Monit Comput. 2022 Aug;36(4):1131-1137. doi: 10.1007/s10877-021-00745-6. Epub 2021 Jul 24. PMID 34302578
- [Background] Debaene B, Frasca D, Moreillon F, D'Hollander AA. 100 Hz-5 s tetanic stimulation to illustrate the presence of "residual paralysis" co-existing with accelerometric 0.90 train-of-four ratio-A proof-of-concept study. Anaesth Crit Care Pain Med. 2021 Aug;40(4):100903. doi: 10.1016/j.accpm.2021.100903. Epub 2021 Jun 17. PMID 34147687
- [Derived] Dubois PE, Moreillon F, Bihin B, De Dorlodot C, Meyer S, Maseri A, Passeraub PA, d'Hollander AA. Spontaneous recovery from rocuronium measured by mechanomyography during 100- or 200-Hz tetanic stimulations compared to normalized train-of-four with acceleromyography. J Clin Monit Comput. 2025 Oct;39(5):1037-1045. doi: 10.1007/s10877-025-01282-2. Epub 2025 Apr 1. PMID 40167977